CLINICAL TRIAL: NCT01445639
Title: Use of Dexmedetomidine for Prophylactic Analgesia and Sedation in Patients After Intracranial Surgery (Prophylactic Analgesia and Sedation Trial, PASTrial)
Brief Title: Dexmedetomidine in Patients After Intracranial Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTH-NICU-2011-02; 2009-03-28 (Other Grant/Funding Number: Beijing Municipal Health Bureau, Beijing, China)
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Central Nervous System Diseases
Keywords: dexmedetomidine; sedation; neurosurgery; postoperative care
MeSH Terms: conditions — Central Nervous System Diseases | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous infusion at rate of 0.4μg/kg/h, during the first 24 hours postoperatively
  Arms: Dexmedetomidine group
Drug: Normal saline — as placebo
  Arms: Placebo group

SUMMARY:
Dexmedetomidine is a highly selective a2-adrenoreceptor agonist that produces dose-dependent sedation and analgesia without respiratory depression. Dexmedetomidine has been used in critically ill medical, surgical, and pediatric patients. No study has been designed specifically to evaluate dexmedetomidine uses in the neurocritical care population. The primary objective is to evaluate the safety and efficacy of dexmedetomidine for prophylactic analgesia and sedation in patients after intracranial surgery.

DETAILED DESCRIPTION:
The PASTrial is a non-commercial, multi-center, randomized, placebo-controlled, double blinded clinical trial. The study compares dexmedetomidine versus normal saline (placebo) in patients after intracranial surgery with delayed extubation. In dexmedetomidine group, infusion (0.4μg/kg/h) is started when patients are admitted to neuro-intensive care unit for postoperative recovery. In control group, patients receive normal saline infusion at the same rate and volume in dexmedetomidine group. The patient's level of sedation is assessed by Sedation-Agitation Scale (SAS) per hour. Midazolam is administered in 0.3-0.5 mg bolus or continuous infusion as SAS above 4. The study is designed primarily to compare the percentage of patients with agitation and requiring midazolam infusion in the 2 study arms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients after intracranial surgery with delayed extubation

Exclusion Criteria:

* emergency operation
* brain stem operation
* preoperative consciousness disorders or epilepsy
* bradycardia, hypotension, acute myocardial infarction, second- or third degree heart block, or need continuous infusions of vasopressor before the start of study drug infusion
* patients enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Mean percentage of hours of optimal sedation. | 24 hours postoperative
  Optimal sedation is defined as SAS score 4.

SECONDARY OUTCOMES:
Percentage of patients with agitation and receiving additional sedatives. | During the first 24 hours postoperatively
  Agitation is defined as SAS above 4. Patients are given midazolam as agitation.

OTHER OUTCOMES:
Percentage of patients with adverse events. | During the first 24 hours postoperatively
  Adverse events include hypotension, bradycardia, airway obstruction, apnea, and consciousness disorders

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Neuro-ICU, Beijing Tiantan Hospital, Capital Medical University
Locations (1):
- Neuro-ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China